CLINICAL TRIAL: NCT03015259
Title: Randomized, Single Blind, Parallel Group, Placebo Controlled, Multidose Study Comparing the Therapeutic Equivalence of a 3M Budesonide/Formoterol Fumarate Inhaler and a Symbicort® Reference Inhaler in Adult Subjects With Asthma
Brief Title: Randomized, Placebo-controlled, Multi-dose, Study Comparing Budesonide/Formoterol to Symbicort® in Asthmatic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kindeva Drug Delivery (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSP-07-000034
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Results first posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-05

CONDITIONS: Asthma
Keywords: bioequivalence
MeSH Terms: conditions — Asthma | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment 1 (Experimental): Generic Budesonide/Formoterol Fumarate Dihydrate (80mcg/4.5mcg) Inhalation Aerosol, two inhalation twice daily, consisting of a 2-week run-in period followed by a 6-week treatment period
  Interventions: Drug: Budesonide/Formoterol fumarate dihydrate
- Treatment 2 (Active Comparator): Symbicort (Budesonide/Formoterol Fumarate Dihydrate) Inhalation Aerosol, two inhalation twice daily, consisting of a 2-week run-in period followed by a 6-week treatment period
  Interventions: Drug: Symbicort
- Treatment 3 (Placebo Comparator): Placebo Inhalation Aerosol, two inhalation twice daily, consisting of a 2-week run-in period followed by a 6-week treatment period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide/Formoterol fumarate dihydrate — Experimental: Treatment 1
  Other Names: Generic Budesonide/Formoterol fumarate dihydrate
  Arms: Treatment 1
Drug: Symbicort — Active Comparator: Treatment 2
  Other Names: Budesonide/Formoterol fumarate dihydrate
  Arms: Treatment 2
Drug: Placebo — Placebo Comparator: Treatment 3
  Arms: Treatment 3

SUMMARY:
A randomized multiple-dose, placebo-controlled, parallel group design consisting of a 2-week run-in period followed by a 6-week treatment period of the placebo, Test product (Budesonide 80 mcg / Formoterol fumarate dihydrate 4.5 mcg), or Reference product Symbicort® inhalation aerosol.

DETAILED DESCRIPTION:
This is a pivotal trial that will examine therapeutic equivalence of a new generic fixed-dose combination product containing Budesonide 80 mcg / Formoterol fumarate dihydrate 4.5 mcg and reference listed drug (RLD) Symbicort® inhalation aerosol in adult patients with chronic but stable asthma as defined in National Asthma Education and Prevention Program Expert Panel Report 3 (NAEPP 3) guidelines. To ensure adequate study sensitivity the test and reference products should both be statistically superior to placebo (p<0.05) with regard to the bioequivalent study primary endpoints.

A secondary study objective is the safety and tolerability of the test compound.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female subjects of non-childbearing or of childbearing potential committed to consistent and correct use of an acceptable method of birth control
* Diagnosed with asthma, as defined by the National Asthma Education and Prevention Program (NAEPP),at least 6 months prior to screening
* Moderate-to-severe asthma with a pre-bronchodilator FEV1 of >45% and <85% of predicted normal, measured at least 6 hours after short-acting β agonist (SABA)and at least 24 hours after the last dose of long-acting β agonist (LABA), at the screening visit and on the day of treatment
* >15% and >0.20 L reversibility of FEV1 within 30 minutes following 360 mcg of albuterol inhalation (pMDI)
* Patients should be stable on their chronic asthma treatment regimen for at least 4 weeks prior to enrollment
* Currently non-smoking; having not used tobacco products (i.e., cigarettes, cigars, pipe tobacco) within the past year, and having < 10 pack-years of historical use
* Able to replace current regularly scheduled short-acting β agonists (SABAs) with salbutamol/albuterol inhaler for use only on an as-needed basis for the duration of the study (subjects should be able to withhold all inhaled SABAs for at least 6 hours prior to lung function assessments on study visits)
* Willing to discontinue their asthma medications (inhaled corticosteroids and long-acting β agonists) during the run-in period and for the remainder of the study
* Willingness to give their written informed consent to participate in the study

Exclusion Criteria:

* Life-threatening asthma, defined as a history of asthma episodes(s) requiring intubation, and/or associated with hypercapnia, respiratory arrest or hypoxic seizures, asthma-related syncopal episodes(s), or hospitalizations within the past year or during the run-in period
* Significant respiratory disease other than asthma (chronic obstructive pulmonary disease (COPD), interstitial lung disease, etc.)
* Evidence or history of clinically significant disease or abnormality including congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, myocardial infarction, or cardiac dysrhythmia. In addition, historical or current evidence of significant hematologic, hepatic, neurologic, psychiatric, renal, or other diseases that, in the opinion of the investigator, would put the patient at risk through study participation, or would affect the study analyses if the disease exacerbated during the study
* Patients who required systemic corticosteroids (for any reason) within the past 4 weeks
* Hypersensitivity to any sympathomimetic drug (e.g., formoterol or albuterol) or any inhaled, intranasal, or systemic corticosteroid therapy
* Patients currently receiving β-blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1762 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: KINDEVA I DD, PhD, Study Chair — Kindeva Drug Delivery
Locations (95):
- United States (95):
  - Clinical Research Center of Alabama LLC, Birmingham, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Clinical Research Consortuim Arizona, Tempe, Arizona
  - Little Rock Allergy and Asthma Clinical Research Center, Little Rock, Arkansas
  - Anaheim Clinical Trials LLC, Anaheim, California
  - Warren W Pleskow MD, Encinitas, California
  - Allergy and Asthma Specialists Medical Group, Huntington Beach, California
  - California Allergy and Asthma Medical Group Inc, Los Angeles, California
  - Jonathan Corren MD, Inc., Los Angeles, California
  - Southern California Institute For Respiratory Diseases, Inc., Los Angeles, California
  - Allergy and Asthma Associates of Southern California, A Medical Group, Inc., Mission Viejo, California
  - Integrated Research Group Inc, Riverside, California
  - Allied Clinical Research LLC, Sacramento, California
  - Allergy and Asthma Associates of Northern California, San Jose, California
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - Allainz Research Institute Inc, Westminster, California
  - Western States Clinical Research Inc, Arvada, Colorado
  - Colorado Allergy and Asthma Centers PC, Centennial, Colorado
  - IMMUNOe Research Centers, Centennial, Colorado
  - Asthma and Allergy Associates PC, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Centers PC, Denver, Colorado
  - Innovative Clinical Research Inc, Lafayette, Colorado
  - Rocky Mountain Center for Clinical Research, Wheat Ridge, Colorado
  - Saint Francis Sleep Allergy and Lung Institute, Clearwater, Florida
  - Southeastern Integrated Medical, Gainesville, Florida
  - Innovative Research of West Florida, Largo, Florida
  - San Marcus Research Clinic Inc, Miami, Florida
  - Prestige Clinical Research Center Inc, Miami, Florida
  - Clintex Research Group, Inc, Miami, Florida
  - Suncoast Research Group LLC, Miami, Florida
  - Applemed Research Inc, Miami, Florida
  - Biotech Pharmaceutical Group, LLC, Miami, Florida
  - Research Institute of South Florida Inc, Miami, Florida
  - Advanced Research Institute Inc, New Port Richey, Florida
  - Emerald Coast Research Associates, Panama City, Florida
  - Allergy and Asthma Dtc, Tallahassee, Florida
  - Asthma and Allergy Center of Chicago Sc, River Forest, Illinois
  - Analab Clinical Research Inc, Lenexa, Kansas
  - Paul Shapero's Private Practice, Bangor, Maine
  - Chesapeake Clinical Research Inc, Baltimore, Maryland
  - Bethesda Allergy Asthma and Research Center LLC, Bethesda, Maryland
  - Genesis Clinical Research and Consulting LLC, Fall River, Massachusetts
  - Infinity Medical Research LLC, North Dartmouth, Massachusetts
  - Northeast Medical Research Associates Inc, North Dartmouth, Massachusetts
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Clinical Research of the Ozarks INC, Columbia, Missouri
  - Clinical Research of the Ozarks Inc, Rolla, Missouri
  - Midwest Clinical Research LLC, St Louis, Missouri
  - The Clinical Research Center LLC, St Louis, Missouri
  - Montana Medical Research, Missoula, Montana
  - Pioneer Clinical Research LLC, Bellevue, Nebraska
  - The Asthma and Allergy Center PC, Bellevue, Nebraska
  - Clinical Research Consortium Nevada, Las Vegas, Nevada
  - Allied Clinical Research LLC, Reno, Nevada
  - Ocean Allergy & Respiratory Research Center, Brick, New Jersey
  - Atlantic Research Center LLC, Ocean Township, New Jersey
  - Princeton Center For Clinical Research, Skillman, New Jersey
  - Allergy Partners of Western North Carolina, Asheville, North Carolina
  - Rapha Institute for Clinical Research, Fayetteville, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Empirical Medical Research, Canton, Ohio
  - Bernstein Clinical Research Center Inc, Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Toledo Center For Clinical Research, Sylvania, Ohio
  - Toledo Institute of Clinical Research, Toledo, Ohio
  - OK Clinical Research, LLC, Edmond, Oklahoma
  - Oklahoma Institute of Allergy and Asthma Clinical Research LLC, Edmond, Oklahoma
  - Santiago Reyes, MD, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute PC, Tulsa, Oklahoma
  - Allergy and Asthma Research Group, Eugene, Oregon
  - Clinical Research Institute of Southern Oregon PC, Medford, Oregon
  - Allergy Associates Research Center LLC, Portland, Oregon
  - Clinical Trial Center LLC, Jenkintown, Pennsylvania
  - Montgomery Medical Inc, Smithfield, Pennsylvania
  - Asthma & Allergy Physicians of Rhode Island Clinical Research Institute, Warwick, Rhode Island
  - ADAC Research, Greenville, South Carolina
  - National Allergy and Asthma Research, LLC, North Charleston, South Carolina
  - S. Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - New Phase Research & Development, Knoxville, Tennessee
  - AARA Research Center, Dallas, Texas
  - Pharmaceutical Research & Consulting Inc, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Metroplex Pulmonology & Sleep Center, McKinney, Texas
  - Central Texas Health Research Corporation, New Braunfels, Texas
  - Quality Assurance Research Center, San Antonio, Texas
  - Allergy and Asthma Research Center PA, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Allergy Asthma Research Institute, Waco, Texas
  - National Clinical Resources Inc, Provo, Utah
  - Timber Lane Allergy and Asthma Research LLC, South Burlington, Vermont
  - Clinical Research Partners LLC, Henrico, Virginia
  - Marycliff Allergy Specialists PS, Spokane, Washington
  - Allergy Asthma and Sinus Center, Greenfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (N=1762) were provided a generic placebo pressurized metered dose inhaler (pMDI) device for use during a 2-week Run-in Period for device training. Then, qualified participants (N=1439) were randomly assigned to treatment on a 3:3:1 ratio of generic budesonide/formoterol fumarate dihydrate, Symbicort, or Placebo, respectively.
Period: Overall Study
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3
Started (Safety Population includes all participants who received at least one dose of a treatment.) | 613 | 622 | 204
Completed (Per Protocol Population includes all participants who provided analyzable data for primary endpoints) | 598 | 604 | 199
Not Completed | 15 | 18 | 5

BASELINE CHARACTERISTICS:
Population: Randomized participants who received at least 1 dose of study drug during Treatment Period
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3 | Total
Number analyzed (Participants) | 613 | 622 | 204 | 1439
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (15.02) | 45.5 (14.44) | 45.5 (14.78) | 45.8 (14.73)
Sex: Female, Male [Count of Participants; unit: Participants] — Randomized participants
  Participants
    Female | 375 | 392 | 137 | 904
    Male | 238 | 230 | 67 | 535
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 153 | 151 | 55 | 359
  Not Hispanic or Latino | 460 | 471 | 149 | 1080
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 5 | 6 | 4 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 107 | 112 | 43 | 262
  White | 490 | 495 | 154 | 1139
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 9 | 3 | 21
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.73 (7.667) | 31.27 (8.108) | 30.93 (7.960) | 30.99 (7.900)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Serial Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 Area calculated over 12 hours (measurements at 0, 1, 2, 3, 4, 6, 8, 12 hours post-dose) on Day 1 of treatment. Because this was a primary endpoint, Per Protocol Population used to calculate this endpoint.
Time Frame: Day 1
Population: Per Protocol Population
Measure: Least Squares Mean (Standard Error); unit: l * hr
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 598 | 604 | 199
l * hr | 4.4453 (0.1552) | 4.2790 (0.1547) | 1.6876 (0.2782)
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2 vs Treatment 3; Only Treatments 1 and 2 were compared for equivalence. Treatment 3 (placebo) was subtracted from both Treatments 1 and 2, as this primary endpoint was baseline adjusted; Test type: Equivalence — To show the clinical equivalence, an analysis of covariance model was fit on the participants from the test budesonide/formoterol fumarate and Symbicort groups, with the endpoint as outcome and treatment, study site and treatment by site interaction as fixed effects and FEV1 baseline value as covariate; Test/Referece LS Mean Ratio = 1.040, 90% CI 2-sided [0.958 to 1.130] — Fieller's formula was applied

2. Primary Outcome: Change From Baseline in FEV1 Measured in the Morning at the End of Treatment Visit
Description: Average predose FEV1 at End of Treatment defined as the average of all predose assessments on Day 42 (+/- 7 days). Baseline was defined as the average of 2 predose FEV1 values obtained on Day 1. The endpoint of baseline-adjusted predose FEV1 at end of treatment was calculated as follows: [FEV1 at end of treatment] - [Baseline FEV1].
Time Frame: Day 1 - Day 49
Population: Per Protocol Population
Measure: Least Squares Mean (Standard Error); unit: liter
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 598 | 604 | 199
liter | 0.3096 (0.0162) | 0.3077 (0.0162) | 0.1236 (0.0285)
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2 vs Treatment 3; Treatments 1 and 2 were baseline adjusted by subtracting Treatment 3 (placebo) from each; Test type: Equivalence — To show the clinical equivalence, an ANCOVA model was fit with the endpoint as outcome and treatment, study site and treatment-by site interaction as fixed effects and FEV1 baseline value as covariate; Test/Reference LS Mean Ratio = 1.004, 90% CI 2-sided [0.889 to 1.140] — Fieller's formula was applied

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants reporting at least one adverse event (safety population)
Time Frame: 6 Weeks
Population: Safety Population: All enrolled participants who received one dose of a treatment drug. This population was larger than the Per Protocol Population that included only those participants who provided analyzable primary endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3
Number analyzed (Participants) | 613 | 622 | 204
Participants
  Upper respiratory tract infection | 12 | 15 | 7
  Nasopharyngitis | 7 | 11 | 4
  Viral upper respiratory tract infection | 6 | 4 | 1
  Bronchitis | 3 | 4 | 2
  Asthma | 17 | 24 | 39
  Cough | 4 | 4 | 3
  Headache | 4 | 8 | 2
  Chest discomfort | 1 | 0 | 2
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2 vs Treatment 3; Comparison of means, no formal statistical comparison; Test type: Other; no statistical significance applied

ADVERSE EVENTS:
Time Frame: Day 1 - Day 70
Description: Subjects who received at least 1 dose during the Treatment Period (Safety Population).
Arm/Group | Treatment 1 | Treatment 2 | Treatment 3
All-Cause Mortality (participants affected / at risk) | 0/613 | 0/622 | 0/204
Serious Adverse Events (participants affected / at risk) | 4/613 | 3/622 | 2/204
Other Adverse Events (participants affected / at risk) | 121/613 | 138/622 | 71/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment 1 (N=613) | Treatment 2 (N=622) | Treatment 3 (N=204)
cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Head injurt (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment 1 (N=613) | Treatment 2 (N=622) | Treatment 3 (N=204)
upper respiratory tract infection (Infections and infestations) | 12 (12) | 15 (15) | 7 (7)
nasopharyngitis (Infections and infestations) | 7 (7) | 11 (11) | 4 (4)
viral upper respiratory tract infection (Infections and infestations) | 6 (7) | 4 (4) | 1 (1)
bronchitis (Infections and infestations) | 3 (3) | 4 (4) | 2 (2)
asthma (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 24 (28) | 39 (48)
cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 3 (3)
gastrointestinal disorders (Gastrointestinal disorders) | 11 (13) | 12 (12) | 2 (4)
injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 8 (8) | 11 (17) | 2 (2)
nervous system disorders (Nervous system disorders) | 9 (12) | 10 (10) | 2 (3)
headache (Nervous system disorders) | 4 (7) | 8 (8) | 2 (3)
infections and infestations (Infections and infestations) | 54 (58) | 58 (61) | 20 (21)
respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 35 (40) | 48 (56) | 48 (64)
musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 8 (11) | 10 (15) | 2 (2)
investigations (Investigations) | 2 (2) | 7 (7) | 3 (3)
general disorders and administration site conditions (General disorders) | 5 (5) | 4 (4) | 2 (3)
chest discomfort (General disorders) | 1 (1) | 0 (0) | 2 (3)
metabolism and nutrition disorders (Investigations) | 4 (4) | 6 (6) | 1 (1)
skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) | 2 (2)
cardia disorders (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
immune system disorders (Immune system disorders) | 2 (2) | 0 (0) | 1 (1)
psychiatric disorders (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
vascular disorders (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
ear and labyrinth disorders (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
eye disorders (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
pregnancy, puerperium, and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
There were no limitations to the trial protocol, no early termination or technical problems.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT03015259/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT03015259/SAP_001.pdf